CLINICAL TRIAL: NCT07220512
Title: The BHFS Study (Better, Harder, Faster, Stronger): Does Neoadjuvant Chemotherapy Improve Fitness for Surgery?
Brief Title: The Better, Harder, Faster, Stronger Study
Status: Recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Atrium Health Wake Forest Baptist (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00129176; ONC-GYN-2401 (Other: Atrium Health Wake Forest Baptist Comprehensive Cancer Center)
Record Dates: First submitted 2025-10-13; First posted 2025-10-24 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Frailty at Older Adults; Ovarian Cancer; Endometrial Cancer; Cognitive Dysfunction; Neoadjuvant Chemotherapy
Keywords: Frailty; ovarian cancer; endometrial cancer; cognitive dysfunction; neoadjuvant chemotherapy
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Cognitive Dysfunction; Frailty | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with ovarian or endometrial carcinoma with planned NACT.: Participants over 55 years old with either ovarian/primary peritoneal/fallopian tube carcinoma or endometrial carcinoma
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — PROs, historical and longitudinal data collection and eFI calculation

SUMMARY:
The purpose of this study is to evaluate changes in the electronic Frailty Index (eFI) score following 3-4 cycles of neoadjuvant chemotherapy (NACT) in participants with advanced ovarian and endometrial cancer.

DETAILED DESCRIPTION:
This observation study is designed investigate changes in frailty and cognitive function in participants with advanced ovarian and endometrial cancer before and after undergoing NACT.

Changes in frailty and cognitive function will be measured using the eFI which is an automated EMR-based tool based that uses a combination of clinical encounters, diagnosis codes, laboratory workups, and Medicare annual wellness visit data as markers of frailty status.

Participants with either ovarian/primary peritoneal/fallopian tube carcinoma or endometrial carcinoma will be approached for interest in participating in this study.

Prior to the first prechemotherapy appointment, eFI will be collected as well as PROs (Functional Assessment of Cancer Therapy - Cognitive Function (FACT-Cog), Patient Health Questionnaire-2 and MoCA (Montreal Cognitive Assessment)) and historical data.

After 3-4 rounds of NACT, eFI, FACT-Cog and MoCA will be collected again. Data on intra-operative and post-operative complications will be collected after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to sign an IRB-approved informed consent.
* Age > 55 years at the time of enrollment.
* Newly diagnosed suspected ovarian/primary peritoneal/fallopian tube carcinoma of any histological subtype, FIGO Stage II-IV, per enrolling investigator, or newly diagnosed suspected endometrial carcinoma of any histologic subtype, FIGO Stage II-IV, per enrolling investigator.
* Planned for 3 or 4 cycles of NACT, with interval cytoreductive surgery planned thereafter.
* Ability to read, understand, and write the English language.
* As determined by the enrolling investigator, ability of the participant to understand and comply with study procedures for the entire length of the study.

Exclusion Criteria:

* History of brain metastases.
* History of poorly controlled psychiatric conditions, defined as hospitalization within the prior 3 months for psychiatric disorders, traumatic brain injury, cerebrovascular event, or dementia, per the enrolling investigator.
* Use of anti-amyloid agents, cholinesterase inhibitors, or glutamate regulators at the time of enrollment.
* Vision impairment that would impede completion of study assessments, per enrolling investigator.

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 55 or older seen in clinic with either ovarian/primary peritoneal/fallopian tube carcinoma or endometrial carcinoma who are planned for NACT
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Change in electronic frailty index (eFI) | From pre- Neoadjuvant Chemotherapy (NACT; no later than 60 days after consent) to post-NACT (no later than 30 days after completion of the last cycle of NACT)
  eFI is an automated electronic medical record-based tool based on a deficit accumulation model of frailty that uses a combination of clinical encounters, diagnosis codes, laboratory workups, and Medicare annual wellness visit data as markers of frailty status.

SECONDARY OUTCOMES:
Change in proportion of participants in the fit/pre-frail (eFI score ≤ 0.21) versus frail category (eFi score > 0.21) | Before and after NACT - At visit 1, no later than 60 days after consent and no later than 30 days after completion of the last cycle of NACT.
  eFI scores are categorized into fit/pre-frail and frail category using the cut of point 0.21
Prevalence of cognitive dysfunction | Before NACT - At visit 1, no later than 60 days after consent
  A MoCA score of 25 or less is used to define cognitive dysfunction
Prevalence of patient-reported cognitive dysfunction | Before NACT - At visit 1, no later than 60 days after consent
  A FACT-Cog PCI score of less than 54 is used to define cognitive dysfunction
Changes in cognitive function as measured by MoCA | Before NACT - At visit 1, no later than 60 days after consent and Post-NACT - no later than 30 days after completion of the last cycle of NACT
  Changes in cognitive function are calculated based on changes in MoCA before and after NACT
Changes in cognitive function as measured by FACT-Cog PCI | Before NACT - At visit 1, no later than 60 days after consent and Post-NACT - no later than 30 days after completion of the last cycle of NACT
  Changes in cognitive function are calculated based on changes in FACT-Cog PCI score before and after NACT
Prevalence of mood disorder | Before NACT - At visit 1, no later than 60 days after consent
  Defined as a PHQ-2 score of 3 or greater

OTHER OUTCOMES:
Length of hospital stay | Post-NACT - no later than 30 days after completion of the last cycle of NACT
  Length of hospital stay
Surgical complication | Post-NACT - no later than 30 days after completion of the last cycle of NACT
  Surgical complication is coded as 0 if no complications occurred, and 1 if any of the complications listed in the NSQIP surgical complication list were present (https://cdn-links.lww.com/permalink/aa/d/aa_2020_05_21_freundlich_aa-d-19-02104r1_sdc1.pdf).
Discharge disposition home vs. rehabilitation facility | Post-NACT - no later than 30 days after completion of the last cycle of NACT
  A binary variable indicating discharge disposition: home (0) vs. rehabilitation facility (1).
Screening rate | at screening
  Screening rate is defined as the proportion of individuals who are potentially eligible, per EMR review, and are willing to be enrolled, out of the total number of participants approached for screening.
Retention rate | Post-NACT - no later than 30 days after completion of the last cycle of NACT
  Retention rate will be defined as the proportion of enrolled participants who completed all required study procedures out of the total number of participants who were initially enrolled.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Kuan-Celarier, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States